CLINICAL TRIAL: NCT04455100
Title: Open-Label, Single-Center, Single-arm, Fixed Sequence Study on the Effect of Itraconazole on the Pharmacokinetics of SHR1459 in Health Subjects
Brief Title: A Phase I Study of SHR1459 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHR1459-I-106
Record Dates: First submitted 2020-06-27; First posted 2020-07-02 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Health, Subjective
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR1459 (Experimental): Following a 10-hour overnight fast, subjects will be administered one dose of SHR1459 orally with 240 mL of ambient temperature water on Day 1. D2-D3 was the cleaning period. Itraconazole will be administered orally 200 mg/time/day form D4 to D8 after meal. On D7 following a 10-hour overnight fast, subjects will be administered SHR1459 and itraconazole 200 mg with 240 mL of ambient temperature water.
  Interventions: Drug: SHR1459/Itraconazole

INTERVENTIONS:
Drug: SHR1459/Itraconazole — SHR1459 will be administered on Day 1 and Day 7. Itraconazole will be administered on Day 4 to Day 8

SUMMARY:
Following a 10-hour overnight fast, subjects will be administered one dose of SHR1459 orally with 240 mL of ambient temperature water on Day 1. D2-D3 was the cleaning period. Itraconazole will be administered orally 200 mg/time/day form D4 to D8 after meal. On D7 following a 10-hour overnight fast, subjects will be administered SHR1459 and itraconazole 200 mg with 240 mL of ambient temperature water.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial and fully understand the content, process and possible adverse of the trial;
2. Able and willing to complete research according to the requirements of the trial;
3. Age at the date of signing informed consent 18 to 55 years old (inclusive), male and female;
4. Male body weight ≥50 kg, female body weight ≥45 kg, body mass index (BMI) between ≥18.0 and ≤26.0 kg/m2, inclusive;
5. Health status: lack of medical history of heart, liver, kidney, digestive tract, nervous system, mental disorders and metabolic abnormalities;
6. Comprehensive physical examination (vital signs, physical examination), routine laboratory examination (blood routine, blood biochemistry, urine routine, etc.), X-chest radiograph, abdominal ultrasound (liver, gallbladder, bile duct, spleen, pancreas, kidney), etc, normal or abnormal and no clinical significance;
7. 12-lead ECG is normal, QTcF for men <430 ms, QTcF for women <450 ms, and heart rate >60;
8. Creatinine clearance (CLCr) ≥80 mL/min, and creatinine is less than or equal to the upper limit of normal value;
9. A negative pregnancy test for females of childbearing potential;
10. Consent to abstinence or use of effective nondrug contraception during the study period and for at least 3 months after the last study drug administration (for women, abstinence or use of effective nondrug contraception during the two weeks prior to study entry is also required).

Exclusion Criteria:

1. Blood donation or loss of more than 200 mL of blood within 1 month of screening; or blood donation or loss of more than 400 mL of blood within 3 months of screening; or received blood
2. Allergic constitution, including severe drug allergy or history of drug allergy; history of allergy to SHR1459, itraconazole, or its accessories;
3. Subject has a history of drug abuse in past 5 years or drug abuse in past 3 months, or is positive for drugs of abuse (eg, morphine/methamphetamine/ketamine/ tetrahydrocannabinolic acid /methylenedioxyethylamphetamine );
4. History of regular alcohol and smoke consumption( exceeding or equal an average weekly intake of 14 standard drinks; 1 drink=150 mL of wine or 360 mL of beer or 45 mL of hard liquor; smoke more than or equal to 5 cigarettes per day)or will not refrain from smoking and drinking during the study;
5. History of cardiovascular dysfunction, myocarditis, coronary heart disease, pathological arrhythmia, stroke and other cardiovascular diseases;
6. Lung diseases, including invasive lung disease, pneumonia, dyspnea, etc;
7. History of chronic kidney disease, renal insufficiency, renal anemia;
8. History of dysphagia or any gastrointestinal disease that affects drug absorption;
9. Any uncontrolled peptic ulcer, colitis, pancreatitis, etc;
10. Had a surgery within 6 months of screening;
11. Important organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and skeletal muscle system (such as uncontrolled diabetes, hypertension, etc.), in the investigator's judgment it is not suitable to participate in this trial;
12. Have taken hepatotoxic drugs for a long period of time (more than 2 consecutive weeks) (such as acetaminophen, statin lipid-lowering drugs, azithromycin, dapsone, clarithromycin, fluconazole, ketoconazole) before the screening;
13. Participated in other clinical trials or used drugs related to this trial within 3 months before screening;
14. Have taken any drugs that alter the activity of liver enzymes 28 days before or during the study;
15. Have taken any prescription or over-the-counter medicine 14 days before study drug administration;
16. Have taken any vitamin products or herbs 14 days before study drug administration;
17. Evidence of clinically significant or other clinical findings show the following diseases (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardio-cerebrovascular diseases);
18. Combine with other viral infections (anti-HCV, anti-HIV positive, HBsAg positive) or syphilis infection;
19. Have ingested grapefruit or products containing grapefruit, dragon fruit, mango, lime, carambola, or food or beverage prepared therefrom 48 hours before taking the study drug;, food or beverage containing caffeine, xanthine or alcohol (Including chocolate, tea, coffee, cola, etc.); strenuous exercise, or other factors that affect the absorption, distribution, metabolism, excretion of drugs, etc;
20. According to the screening chest X-ray and abdominal ultrasound (liver, gallbladder, bile duct, spleen, pancreas, kidney) examination items confirmed abnormal and clinically significant;
21. Vaccination recipients within 4 weeks before screening;
22. Cannot tolerate venous puncture or have a history of halo acupuncture;
23. Lactose intolerant;
24. Required special dietary and refuse the unified diet;
25. Subjects with acute illness from screening to pre-dose;
26. In the investigator's judgment subjects are not suitable to participate in this trial;

    In addition to the above requirements, female volunteers who meet the following conditions should also be excluded:
27. Have taken contraceptives within 30 days before screening (interview);
28. Used long-acting estrogen or progesterone injections (including progesterone intrauterine devices) or implants within 6 months before screening;
29. Subjects had unprotected sex with their partner within 14 days before screening;
30. Female subjects are during in period of lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2020-08-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of SHR1459 | from Day 1 to Day 9
  Peak Plasma Concentration (Cmax) of SHR1459
Pharmacokinetics parameter: AUC of SHR1459 | from Day 1 to Day 9
  Area under the plasma concentration versus time curve (AUC) of SHR1459

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of SHR1459 | from Day 1 to Day 9
  Time of maximum observed concentration (Tmax) of SHR1459
Pharmacokinetics parameter: T1/2 of SHR1459 | from Day 1 to Day 9
  Half time (T1/2) of SHR1459
Pharmacokinetics parameter: CL/F of SHR1459 | from Day 1 to Day 9
  Apparent clearance of SHR1459
Pharmacokinetics parameter: Vz/F of SHR1459 | from Day 1 to Day 9
  Apparent volume of distribution of SHR1459

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided